CLINICAL TRIAL: NCT05968417
Title: Investigation of the Activity of Novel Compounds for the Treatment of Myeloma and Mechanisms of Drug Resistance to Current Therapies
Brief Title: Myeloma Novel Drug Discovery Ver 1.2
Acronym: DISCO
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5106
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with a diagnosis, or suspected diagnosis, of myeloma or related plasma cell disorder: Participants who are undergoing peripheral blood or bone marrow aspirate sampling for diagnostic, staging or follow-up purposes, before, whilst or after receiving anti-myeloma treatment will be approached to collect additional samples for research.
  Interventions: Other: Observational study - sample collection only.

INTERVENTIONS:
Other: Observational study - sample collection only. — No intervention - blood and/or bone marrow sample collection only

SUMMARY:
Myeloma is a bone marrow cancer with over 5000 patients diagnosed in the UK each year. Researchers are committed to improving understanding of myeloma and developing more effective treatments with fewer side effects in order to improve patient outcomes. In order to do this, researchers are collecting samples of blood and bone marrow to test the activity of potential new treatments in the laboratory and to understand what may be the cause of some treatments not working.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have a diagnosis, or suspected diagnosis, of myeloma or related plasma cell disorder
2. Participants who are undergoing a peripheral blood or bone marrow aspirate sampling for diagnostic, staging or follow-up purposes, before, whilst or after receiving anti-myeloma treatment
3. Participants aged 18 years of age or above
4. Participants willing to consent to an additional sample being taken at the time of their peripheral blood or bone marrow aspirate sampling

Exclusion Criteria:

1. Participants unable to provide consent
2. Participants with known active infectious diseases (e.g. HIV, Hepatitis B/C, COVID) that pose a risk to the use of the sample in the laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have a diagnosis, or suspected diagnosis, of myeloma or related plasma cell disorder
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2033-02-28 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Cell viability | 12 months
  Myeloma cell viability when incubated with standard of care and novel compounds.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom